CLINICAL TRIAL: NCT02414555
Title: Perioperative Fluid Management in Patients Receiving Major Abdominal Surgery - Effects of Normal Saline Versus an Acetate Buffered Balanced Infusion Solution on the Necessity of Catecholamines for Cardiocirculatory Support, a Randomized Controlled Double-blind Trial
Brief Title: Perioperative Fluid Management in Patients Receiving Major Abdominal Surgery - Effects of Normal Saline Versus an Acetate Buffered Balanced Infusion Solution on the Necessity of Catecholamines for Cardiocirculatory Support
Acronym: KATECHOL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Patient Safety
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Pfortmueller Carmen Andrea, Department of Anesthesiology, Intensive Care and Pain Management, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: v1.104112014
Record Dates: First submitted 2015-03-23; First posted 2015-04-10 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Critical Illness
Keywords: Fluid Management
MeSH Terms: conditions — Critical Illness | interventions — Vasoconstrictor Agents; Phenylephrine; Norepinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaCl 0.9% BBraun (normale saline) (Active Comparator): 154mmol/l sodium, 154mmol/l chloride
  Interventions: Drug: vasopressor; Drug: fluid bolus; Device: oesophagus doppler (CardioQ); Drug: Normal Saline; Device: arterial cannulation; Device: intravenous peripheral line insertion (17 gauge)
- Elo-Mel Isoton (balanced acetat-based infusate) (Active Comparator): sodium 140mmol/l, potassium 5.0mmol/l, calcium 2.5mmol/l, magnesium 1.5mmol/l, chlorid 108mmol/l, acetate 45mmol/l
  Interventions: Drug: vasopressor; Drug: fluid bolus; Device: oesophagus doppler (CardioQ); Device: arterial cannulation; Device: intravenous peripheral line insertion (17 gauge); Drug: Elo-Mel Isoton (balanced acetat-based infusate)

INTERVENTIONS:
Drug: vasopressor — Patients receive oesophageal doppler-based hemodynamic support either with fluid or with vasopressor
  Other Names: phenylephrine, norepinephrine
Drug: fluid bolus
Device: oesophagus doppler (CardioQ)
Drug: Normal Saline
  Arms: NaCl 0.9% BBraun (normale saline)
Device: arterial cannulation
Device: intravenous peripheral line insertion (17 gauge) — for fluid bolus administration
Drug: Elo-Mel Isoton (balanced acetat-based infusate)
  Arms: Elo-Mel Isoton (balanced acetat-based infusate)

SUMMARY:
Background Intraoperative hypotension is a common problem that significantly contributes to perioperative mortality and morbidity. At the moment the "gold standard" for perioperative fluid management is the so called "goal-directed therapy" that features fluid resuscitation followed if necessary catecholamines if needed for perioperative cardiocirculatory support.

Worldwide the so called "physiological" sodium chlorid (0.9% NaCl) solution is the most often used infusate for perioperative fluid management. Despite its widespread use physiological saline has its major disadvantages such as the increased incidence of metabolic acidosis. Nevertheless catecholamines have their significant side effects as well (eg diminished renal perfusion, increased cardiovascular morbidity) and they therefore should be used with caution.

In a prior study by group members on patients undergoing renal transplantation receiving either physiological saline or an acetate-buffered infusate showed a 50% decrease in catecholamine necessity in the acetate-buffered infusate group. The investigators therefore would like to evaluate the effects of the perioperative fluid choice on the necessity of catecholamine use.

Aim

* Evaluation of the perioperative fluid choice on the necessity of catecholamines for cardiocirculatory support.
* Description of the relationship between perioperative fluid choice and minimal blood pressure as well as the time to catecholamine use and their dosage.

Methods The investigators plan a prospective randomized-controlled trial of all patients undergoing major abdominal surgery at the Vienna General Hospital and Medical University of Vienna. Fluid management and catecholamine use will be based on a oesophageal Doppler -based treatment scheme.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for open elective major abdominal surgery and expected to last a minimum of 2 hours will be included in the study.

(Major abdominal surgery includes all gynecological, urological and general surgical operations requiring laparotomy)

Exclusion Criteria:

* Patients younger than 18 years of age
* Patients unable to give informed consent
* Pregnancy or breastfeeding
* Patients transferred form the intensive care unit to the operating theater
* Patients with an already established catecholamine therapy
* Emergency operation
* Chronic inflammatory diseases (chronic inflammatory rheumatoid diseases, chronic inflammatory renal diseases, chronic inflammatory infectious diseases, chronic inflammatory bowel diseases, chronic liver disease with signs of liver insufficiency)
* Severe cardiovascular disease (heart disease with an ejection fraction below 30%, instable coronary syndromes, severe valvular disease)
* Any signs of infection or sepsis
* Any contraindication for oesophageal Doppler monitoring (oesophageal and aortic pathology, planned oesophageal resection)
* Renal insufficiency with a glomerular filtration rate below 30ml/min
* Patients with additional epidural anesthesia are excluded from the study if epidural anesthesia is planned to be used for analgesia intraoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
catecholamine use to maintain target mean arterial pressure | hours of anesthesia (max 10 hours)

SECONDARY OUTCOMES:
difference in dose of catecholamines to maintain cardiovascular stability | hours of anesthesia (max 10 hours)
difference in volume to maintain cardiovascular stability | hours of anesthesia (max 10 hours)
unplanned ICU transfers | hours of anesthesia (max 10 hours)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Markstaller, MD, Study Director — Clinic for General Anesthesia, Intensive Care and Pain Management, Medical University of Vienna, Vienna, Austria
Locations (1):
- Department of General Anesthesiology, Intensive Care and Pain Management, Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pfortmueller CA, Funk GC, Reiterer C, Schrott A, Zotti O, Kabon B, Fleischmann E, Lindner G. Normal saline versus a balanced crystalloid for goal-directed perioperative fluid therapy in major abdominal surgery: a double-blind randomised controlled study. Br J Anaesth. 2018 Feb;120(2):274-283. doi: 10.1016/j.bja.2017.11.088. Epub 2017 Dec 2. PMID 29406176